CLINICAL TRIAL: NCT01223456
Title: A Descriptive Study of the Efficacy and Safety of ONGLYZA (Saxagliptin) Under Conditions of Actual Use in the Philippines
Brief Title: Safety and Efficacy Study of ONGLYZA (Saxagliptin) Under Conditions of Actual Use
Acronym: ONGLYZA PMS
Status: Terminated | Type: Observational
Why Stopped: Inability to recruit adequate number of patients within the specified time period.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CPH-DUM-2010/1
Record Dates: First submitted 2010-10-14; First posted 2010-10-19 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Saxagliptin; type 2 diabetes; clinical practice
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This post marketing surveillance study aims to monitor the safety and efficacy of ONGLYZA under conditions of actual use in patients who are diagnosed with diabetes mellitus type 2 and are prescribed ONGLYZA by their physician.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 2 Diabetes Mellitus
* Prescribed Saxagliptin by patient's attending physician

Exclusion Criteria:

* Known allergic or serious adverse reaction to Saxagliptin
* Pregnant or breastfeeding patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: several private and government hospitals
Sampling Method: Non-Probability Sample
Enrollment: 542 (Actual)
Dates: Start 2010-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Adverse events observed during the treatment duration | Upon enrollment and initiation of Saxagliptin up to 14 days post follow-up
Clinical Response determined by cure rate | Up to three (3) months after initiation of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Milagros Tan, MD, Study Director — AstraZeneca Philippines; Emmanuel Arca, MD, Study Chair — AstraZeneca Philippines
Locations (11):
- Philippines (11):
  - Research Site, Batangas, Batangas
  - Research Site, Cebu City, Cebu
  - Research Site, Davao City, Davao Region
  - Research Site, Iloilo City, Iloilo
  - Research Site, Las Piñas, Manila
  - Research Site, Makati, Manila
  - Research Site, Manila, Manila
  - Research Site, Pasig, Manila
  - Research Site, Quezon City, Manila
  - Research Site, Mabalacat, Pampanga
  - Research Site, Manila